CLINICAL TRIAL: NCT05046249
Title: Swiss Chiropractic Cohort (Swiss ChiCo) Study: A Nationwide Practice-Based Research Network Project
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other); University of Southern Denmark, Department of Sports Science and Clinical Biomechanics (Unknown); Swiss Chiropractic Association (ChiroSuisse) (Unknown); Swiss Chiropractic Patient Association (Pro Chiropractic Switzerland) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SwissChiCo-PBRN
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Pain
Keywords: Chiropractic; Health care quality; Musculoskeletal health; Manual medicine
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chiropractic clinicians: Swiss chiropractic clinicians

SUMMARY:
The Swiss chiropractic cohort (Swiss ChiCo) practice-based research network (PBRN) is nationwide research project with the aim to develop a musculoskeletal focused PBRN within the Swiss chiropractic setting and describe the characteristics of clinicians recruited. Development of the PBRN has been guided through participatory engagement of multiple stakeholders including patients, clinicians, scientists, and policymakers.

DETAILED DESCRIPTION:
Management of musculoskeletal (MSK) conditions is moving away from traditional medical treatments such as pain medication and towards more physical and preventative approaches. As a result, there is a need to describe manual care approaches to make informed decisions on how best to use this capacity in the current health care system. While this literature is emerging, very little is collected from clinical settings where the large majority of MSK care occurs. The lack of clinically collected data creates gaps in patient-centred research and difficulties with knowledge implementation in treatment settings.

To help bridge this divide, countries such as the United Kingdom, Canada, Sweden, and Australia have established MSK-focused practice-based research networks (PBRNs). PBRNs are sustained collaborations between practitioners and academicians. This collaboration allows patient recruitment from diverse clinical settings and allows practitioners to be more actively involved in the research process. As a result data collected, and subsequent recommendations may have greater clinical utility than that which comes from more traditional research-only settings.

This study aims to develop a MSK focused PBRN within the Swiss chiropractic setting and describe the characteristics of clinicians recruited. It represents a collaborative effort of international researchers, Swiss chiropractic clinicians, and the chiropractic patient and clinical associations in Switzerland (Pro Chiropractic Switzerland and ChiroSuisse). Clinicians will endorse participation in the PBRN by completing an electronic study form. Once established, nested sub-studies will be conducted within this new clinical research environment. Through stakeholder engagement and institutional support, the Swiss ChiCo PBRN can serve as an important resource to advance chiropractic and MSK health services research.

ELIGIBILITY:
Inclusion Criteria:

* Active clinician members of the Swiss Chiropractic Association (ChiroSuisse)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All active chiropractors in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Self-confidence in clinical management of patients with low back pain | Baseline
  Assessment via practitioner self-confidence scale (PCS, 4-20). The PCS contains four items with a total score of 20 where 4 represents greatest self-confidence and 20 represents the lowest self-confidence towards clinical management of patients with low back pain.
Biomedical versus biopsychosocial treatment orientation | Baseline
  Assessment via pain attitudes and beliefs scale musculoskeletal version (PABS-MSK). The PABS-MSK contains two domains, a higher score on the biomedical domain (PABS-MSK-BM, score range 10-60) represents a higher biomedical orientation. A higher score on the biopsychosocial domain (PABS-MSK-BPS, score range 10-60) represents a higher biopsychosocial orientation.
Participation proportion (feasibility outcome) | Baseline
  Proportion of eligible clinicians who participate
Motivation for clinician participation in a PBRN sub-study (feasibility outcome) | Baseline
  Assessment via visual analog scale (VAS, 0-100). A higher score reflects higher motivation for clinician participation in a PBRN sub-study.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Hincapié, DC PhD, Principal Investigator — Balgrist University Hospital and University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data may be made available for research purposes. Requests, including a synopsis of the study plan, can be addressed to the central contact person.

REFERENCES:
- [Background] Lalji R, Hofstetter L, Kongsted A, von Wyl V, Puhan MA, Hincapie CA. Swiss chiropractic practice-based research network and musculoskeletal pain cohort pilot study: protocol of a nationwide resource to advance musculoskeletal health services research. BMJ Open. 2022 Jul 13;12(7):e059380. doi: 10.1136/bmjopen-2021-059380. PMID 35831057
- [Result] Lalji R, Hofstetter L, Kongsted A, von Wyl V, Puhan MA, Hincapie CA. The Swiss chiropractic practice-based research network: a population-based cross-sectional study to inform future musculoskeletal research. Sci Rep. 2023 Apr 6;13(1):5655. doi: 10.1038/s41598-023-32437-3. PMID 37024506
- See also: Musculoskeletal Epidemiology Research Group, Balgrist University Hospital, Project webpage — https://www.balgrist.ch/en/research/research-units/research-orthopaedics/musculoskeletal-epidemiology-research/research-projects/